CLINICAL TRIAL: NCT04272359
Title: Prospective, Parallel Goups Study, Aimed to Evaluating Possible Benefits of the Treatment of New Generation Hypoglycaemic Drugs Compared to Sulphonylureas for the Tratment of Type 2 Diabetes Mellitus
Brief Title: Substitution of Sulfonylureas With New Generation of Hypoglycemic Drugs for the Treatment of Type 2 Diabetes Mellitus
Acronym: Sulfa-Zero
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Clinical Professor, University of Milan
Other Study IDs: Sacco Milan
Record Dates: First submitted 2019-10-30; First posted 2020-02-17 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Diet, Healthy; Renal Function Disorder; Albuminuria
Keywords: Sulfaniluree/glinidi
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: SGLT2 inibitori +/- Metformin
  Interventions: Drug: Sulfa-zero: possible benefits of the treatment of new generation hypoglycaemic drugs compared to sulphonylureas
- Group 2: DPP4 inibitori +/- Metformin
  Interventions: Drug: Sulfa-zero: possible benefits of the treatment of new generation hypoglycaemic drugs compared to sulphonylureas
- Group 3: GLP1-RA + Long-Acting Insulin +/- Metformin
  Interventions: Drug: Sulfa-zero: possible benefits of the treatment of new generation hypoglycaemic drugs compared to sulphonylureas
- Group 4: SGLT2 inibitori + DPP4 inibitori +/- Metformin
  Interventions: Drug: Sulfa-zero: possible benefits of the treatment of new generation hypoglycaemic drugs compared to sulphonylureas

INTERVENTIONS:
Drug: Sulfa-zero: possible benefits of the treatment of new generation hypoglycaemic drugs compared to sulphonylureas — Substitution of sulfonylureas with other classes of new hypoglycaemic drugs. In every group, it will be evaluated:
  * efficacy in terms of glycometabolic compensation (glycemia, HbA1c, lipid profile);
  * effects on BMI, blood pressure monitoring and hypoglycemic risk;
  * changes in renal function and microalbuminuria;
  * tolerability and side effects of the new therapeutic regimes;
  * therapeutic adherence;
  * post-prandial glycemic excursion, determined by a 6-point glycemic diary (pre- and 2h post-prandial glucose values) to be performed at home in the week before the scheduled follow-up visit;
  * effects on chronic complications of diabetes and cardiovascular safety.
  Other Names: Shift to new generation therapeutic regimens

SUMMARY:
This is a multicentric, prospective, parallel groups study. Patient recruitment will be carried out at the U.O. Departmental Endocrinology and Diabetology ASST FBF Sacco, Fatebenefratelli and Ophthalmic Hospital, and at the SSD of Endocrine Diseases and Diabetology ASST FBF Sacco, L. Sacco Hospital.

At the screening visit, patients being treated with sulfonylureas / glinids will be shifted, depending on the subject's biochemical and phenotypic characteristics, based on current prescribing criteria and diabetes complications, to one of 4 different types of treatment:

1. GROUP 1: SGLT2 inhibitors +/- Metformin
2. GROUP 2: DPP4 inhibitors +/- Metformin
3. GROUP 3: GLP1-RA + Long-acting insulin +/- Metformin
4. GROUP 4: SGLT2 inhibitors + DPP4 inhibitors +/- Metformin At the screening visit the clinician will evaluate which new treatment to assign to the patient, based on the subject's biochemical and phenotypic characteristics, current prescribing criteria and existing complications (Algorithm for the treatment of diabetes mellitus, SID-AMD Care Standard 2018)

DETAILED DESCRIPTION:
Approximately 500 T2DM patients aged ≥18 years will be enrolled according to the guidelines of the American Diabetes Association (ADA) with poor glycemic control (hemoglobin A1c [A1C] ≥6.5% and ≤11% [≥58 mmol / mol and ≤97 mmol / mol]), in stabilized treatment with sulfonylureas / glinids, which meet all the study enrollment criteria.

During the study 7 visits are scheduled which coincide with the routine diabetic visits.

During the scheduled visits the patients of the study will be subjected to:

* Enrollment on the first visit if the inclusion criteria are met and those of exclusion are absent
* Anamnestic and clinical collection
* Evaluation of the type of treatment to which they have been assigned and possible modification of drug therapy in the in case that the desired glycemic target has not yet been reached up.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* 6.5% <HbA1c <11%;
* Diagnosis of type 2 diabetes mellitus;
* Active treatment with sulfonylureas / glinids, both in monotherapy and in association with other long-acting hypoglycemic / insulins.
* Written informed consent of the patient or a legal guardian signed and dated

Exclusion Criteria:

* Patients suffering from severe systemic diseases, fever, known chronic inflammatory states
* PCR determinants> 10 mg/L;
* HbA1c> 11% or HbA1c <6.5%;
* Use of corticosteroids at the time of enrollment;
* Poor patient understanding of spoken and written Italian;
* Absent compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The size of the sample chosen is such in consideration of the average number of patients suffering from type 2 Diabetes Mellitus treated by the Diabetology Clinics of the participating structures in the study and therefore will allow us to complete enrollment within the first months of the study
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-10-06 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of the glyco-metabolic parameters | 12 months
  Evaluation of the new generation hypoglicemic drugs on Hba1c, blood glucose, lipidic profile
Therapeutic adherence | 12 months
  Assessment of adherence to the doctor's prescription of new generation hypoglycaemic drugs
Long-term diabetes complications | 12 months
  Evaluation of the effect of new generation hypoglycemic drugs on the long-term complications of diabetes compared to the effect obtained with sulphonylureas

SECONDARY OUTCOMES:
Values of the insulin-sensitivity | 12 months
  Evaluation of the effect of new generation hypoglycemic drugs on the insulin secretion of diabetes compared to the effect obtained with sulphonylureas.
Therapeutic compliance, even in populations over 70 years. | 12 months
  Evaluation of the effect of new generation hypoglycemic drugs on therapeutic adherence with respect to the effect obtained with sulphonylureas even in older subjects.
Insulin parameters after shift to new-generation hypoglycaemic therapeutic regimens | 12 months
  HOMA-IR and HOMA-B% insulin parameters evaluation in patients not in insulin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fiorina, MD, PhD, Principal Investigator — University of Milan
Locations (1):
- ASST FBF-Sacco P.O. Sacco/Fatebenefratelli e Oftalmico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garber A, Henry R, Ratner R, Garcia-Hernandez PA, Rodriguez-Pattzi H, Olvera-Alvarez I, Hale PM, Zdravkovic M, Bode B; LEAD-3 (Mono) Study Group. Liraglutide versus glimepiride monotherapy for type 2 diabetes (LEAD-3 Mono): a randomised, 52-week, phase III, double-blind, parallel-treatment trial. Lancet. 2009 Feb 7;373(9662):473-81. doi: 10.1016/S0140-6736(08)61246-5. Epub 2008 Sep 24. PMID 18819705
- [Background] Kahn SE, Haffner SM, Heise MA, Herman WH, Holman RR, Jones NP, Kravitz BG, Lachin JM, O'Neill MC, Zinman B, Viberti G; ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med. 2006 Dec 7;355(23):2427-43. doi: 10.1056/NEJMoa066224. Epub 2006 Dec 4. PMID 17145742
- [Background] Zhang Y, Hong J, Chi J, Gu W, Ning G, Wang W. Head-to-head comparison of dipeptidyl peptidase-IV inhibitors and sulfonylureas - a meta-analysis from randomized clinical trials. Diabetes Metab Res Rev. 2014 Mar;30(3):241-56. doi: 10.1002/dmrr.2482. PMID 24123720
- [Background] Charbonnel B, Schernthaner G, Brunetti P, Matthews DR, Urquhart R, Tan MH, Hanefeld M. Long-term efficacy and tolerability of add-on pioglitazone therapy to failing monotherapy compared with addition of gliclazide or metformin in patients with type 2 diabetes. Diabetologia. 2005 Jun;48(6):1093-104. doi: 10.1007/s00125-005-1751-1. Epub 2005 May 12. PMID 15889234
- [Background] Matthews DR, Charbonnel BH, Hanefeld M, Brunetti P, Schernthaner G. Long-term therapy with addition of pioglitazone to metformin compared with the addition of gliclazide to metformin in patients with type 2 diabetes: a randomized, comparative study. Diabetes Metab Res Rev. 2005 Mar-Apr;21(2):167-74. doi: 10.1002/dmrr.478. PMID 15386821
- [Background] Nauck M, Frid A, Hermansen K, Thomsen AB, During M, Shah N, Tankova T, Mitha I, Matthews DR. Long-term efficacy and safety comparison of liraglutide, glimepiride and placebo, all in combination with metformin in type 2 diabetes: 2-year results from the LEAD-2 study. Diabetes Obes Metab. 2013 Mar;15(3):204-12. doi: 10.1111/dom.12012. Epub 2012 Oct 11. PMID 22985213
- [Background] Cefalu WT, Leiter LA, Yoon KH, Arias P, Niskanen L, Xie J, Balis DA, Canovatchel W, Meininger G. Efficacy and safety of canagliflozin versus glimepiride in patients with type 2 diabetes inadequately controlled with metformin (CANTATA-SU): 52 week results from a randomised, double-blind, phase 3 non-inferiority trial. Lancet. 2013 Sep 14;382(9896):941-50. doi: 10.1016/S0140-6736(13)60683-2. Epub 2013 Jul 12. PMID 23850055
- [Background] Nauck MA. Incretin-based therapies for type 2 diabetes mellitus: properties, functions, and clinical implications. Am J Med. 2011 Jan;124(1 Suppl):S3-18. doi: 10.1016/j.amjmed.2010.11.002. PMID 21194578
- [Background] Del Prato S, Nauck M, Duran-Garcia S, Maffei L, Rohwedder K, Theuerkauf A, Parikh S. Long-term glycaemic response and tolerability of dapagliflozin versus a sulphonylurea as add-on therapy to metformin in patients with type 2 diabetes: 4-year data. Diabetes Obes Metab. 2015 Jun;17(6):581-590. doi: 10.1111/dom.12459. Epub 2015 Apr 6. PMID 25735400
- [Background] Nauck MA. Update on developments with SGLT2 inhibitors in the management of type 2 diabetes. Drug Des Devel Ther. 2014 Sep 11;8:1335-80. doi: 10.2147/DDDT.S50773. eCollection 2014. PMID 25246775
- [Background] Ridderstrale M, Andersen KR, Zeller C, Kim G, Woerle HJ, Broedl UC; EMPA-REG H2H-SU trial investigators. Comparison of empagliflozin and glimepiride as add-on to metformin in patients with type 2 diabetes: a 104-week randomised, active-controlled, double-blind, phase 3 trial. Lancet Diabetes Endocrinol. 2014 Sep;2(9):691-700. doi: 10.1016/S2213-8587(14)70120-2. Epub 2014 Jun 16. PMID 24948511
- [Background] Maedler K, Carr RD, Bosco D, Zuellig RA, Berney T, Donath MY. Sulfonylurea induced beta-cell apoptosis in cultured human islets. J Clin Endocrinol Metab. 2005 Jan;90(1):501-6. doi: 10.1210/jc.2004-0699. Epub 2004 Oct 13. PMID 15483097
- [Background] Karl DM, Gill J, Zhou R, Riddle MC. Clinical predictors of risk of hypoglycaemia during addition and titration of insulin glargine for type 2 diabetes mellitus. Diabetes Obes Metab. 2013 Jul;15(7):622-8. doi: 10.1111/dom.12072. Epub 2013 Feb 24. PMID 23350795
- [Background] Holstein A, Plaschke A, Egberts EH. Lower incidence of severe hypoglycaemia in patients with type 2 diabetes treated with glimepiride versus glibenclamide. Diabetes Metab Res Rev. 2001 Nov-Dec;17(6):467-73. doi: 10.1002/dmrr.235. PMID 11757083
- [Background] A study of the effects of hypoglycemia agents on vascular complications in patients with adult-onset diabetes. VI. Supplementary report on nonfatal events in patients treated with tolbutamide. Diabetes. 1976 Dec;25(12):1129-53. doi: 10.2337/diab.25.12.1129. No abstract available. PMID 992232
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Nunes AP, Iglay K, Radican L, Engel SS, Yang J, Doherty MC, Dore DD. Hypoglycaemia seriousness and weight gain as determinants of cardiovascular disease outcomes among sulfonylurea users. Diabetes Obes Metab. 2017 Oct;19(10):1425-1435. doi: 10.1111/dom.13000. Epub 2017 Jul 21. PMID 28497592
- [Background] Middleton TL, Wong J, Molyneaux L, Brooks BA, Yue DK, Twigg SM, Wu T. Cardiac Effects of Sulfonylurea-Related Hypoglycemia. Diabetes Care. 2017 May;40(5):663-670. doi: 10.2337/dc16-1972. Epub 2017 Feb 21. PMID 28223296